CLINICAL TRIAL: NCT05303428
Title: Study of Low-intensity Focused Ultrasound Effects on Cognitive fMRI Signals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Wynn Legon, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22-243
Record Dates: First submitted 2022-03-04; First posted 2022-03-31 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Cognitive Change

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LIFU, fMRI Cognitive (Experimental): fMRI resting and cognitive tasks performed after LIFU application to known brain region of interest or active sham region (within participant all conditions tested).
  Interventions: Other: Neuromodulation with low-intensity focused ultrasound

INTERVENTIONS:
Other: Neuromodulation with low-intensity focused ultrasound — application of LIFU to induce temporary neuromodulation, effects tested with resting state and task based fMRI scanning.

SUMMARY:
Study aims to examine the effects of noninvasive brain stimulation on brain signals. This insight may have potential clinical implications for addiction, pain, and mental health populations. Participants will receive MRI and CT imaging. Participants receive low-intensity focused ultrasound (LIFU) to temporarily change brain activity. Participants then receive fMRI scans to measure changes in both resting and cognitive brain signaling using structured tasks. Heart rate, blood pressure, respiratory rate, and skin moisture is monitored. Participants complete a battery of questionnaires, both behavioral and symptom monitoring. The study takes place over 4 study visits.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, all ethnicities, who understand and speak English.

Exclusion Criteria:

1. Claustrophobia (scanning environment may be uncomfortable).
2. Contraindications to MRI: including pacemaker, aneurysm clips, neurostimulators, cochlear implants, metal in eyes, steel worker, or other implants.
3. Contraindications to CT: pregnancy
4. Active medical disorder or treatment with potential CNS effects (e.g. Alzheimer's)
5. History of neurologic disorder. (e.g. Parkinson's, Epilepsy, or Essential Tremor)
6. History of head injury resulting in loss of consciousness for >10 minutes.
7. History of alcohol or drug dependence (through self-report).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-10 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
fMRI Signals - Cognition | Participant study duration, approximately 3 weeks.
  Changes in fMRI signals of region of interest during a cognitive task

SECONDARY OUTCOMES:
Executive function task performance | Participant study duration, approximately 3 weeks.
  Testing effects of LIFU on altered task performance

OTHER OUTCOMES:
Assess for changes in physiological measures | Participant study duration, approximately 3 weeks.
  Monitoring for any changes in heartrate, blood pressure, respiratory rate, or galvanic skin response throughout testing

IPD SHARING:
Plan to Share IPD: No